CLINICAL TRIAL: NCT00879671
Title: Effects of Lutein Supplementation on Macular Pigment Optical Density and Visual Acuity in Patients With Age-related Macular Degeneration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. Priv.-Doz., Medical University of Vienna
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OPHT-100205
Record Dates: First submitted 2009-04-09; First posted 2009-04-10 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Age-Related Macular Degeneration
Keywords: lutein; nonexudative AMD; MPOD; Supplementary Concepts
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Lutamax
  Interventions: Dietary Supplement: lutamax (leutein)
- 2 (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: lutamax (leutein) — leutein 20 mg for 3 months, then lutein 10 mg
  Arms: 1
Dietary Supplement: placebo — Placebo capsules identical in taste and appearance
  Arms: 2

SUMMARY:
The macular pigment (MP) in humans consists of the yellow, blue-absorbing carotenoids lutein and zeaxanthin. The highest concentrations of lutein and zeaxanthin are found in the fovea. Since light entering the eye passes through the MP before reaching the photo receptors it absorbs a significant portion of short-wavelength light. There is evidence that this absorbing properties of the MP as well as the ability of inactivating highly reactive oxygen species are protective for the retina.

Age-related macular degeneration is the leading cause of blindness among developed countries. The pathogenesis of this disease remains unknown. There is, however, evidence that low fruit and vegetable consumption increases the risk of Age-Related Macular Degeneration (AMD). Accordingly, it has been hypothesized that lutein supplementation may be beneficial in AMD. The present study investigates whether 6 months lutein supplementation increases MP optical density (OD), influences visual acuity, depth and dimension of central scotoma and alters symptoms in patients with AMD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with nonexudative AMD (either categories 2, 3 or 4 according to the AREDS criteria; in group 4 the eyes with no-advanced AMD will be included, Age-Related Eye Disease Study Research Group 2001)
* Age between 50 and 90 years
* Clear non-lenticular ocular media
* Visual acuity > 0.4

Exclusion Criteria:

* Primary retinal pigment epithelium atrophy > 125 µm
* Moderate or severe non-proliferative diabetic retinopathy, proliferative diabetic retinopathy
* Participation in a clinical trial in the 3 weeks preceding the study
* Previous treatment with lutein within 3 month of study initiation
* History of hypersensitivity to the trial drug or to drugs with a similar chemical structure
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with, distribution, metabolism or excretion of study drugs
* Ocular surgery within the last 6 months
* Treatment with photosensitizing drugs

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2006-11; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Macular pigment optical density (MPOD) as measured with optical reflectometry | 5 minutes

SECONDARY OUTCOMES:
Visual acuity using ETDRS charts | 15 minutes
Central visual field defects assessed with scanning laser scotometry | 30 minutes
Changes in fundus appearance as documented with fundus photos | 5 minutes
Determination of an increased systemic antioxidative state in plasma and low density lipoprotein and Plasma lutein concentrations | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Schmidt-Erfurth, Prof. Dr., Principal Investigator — Department of Opthalmology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Evans JR, Lawrenson JG. Antioxidant vitamin and mineral supplements for slowing the progression of age-related macular degeneration. Cochrane Database Syst Rev. 2023 Sep 13;9(9):CD000254. doi: 10.1002/14651858.CD000254.pub5. PMID 37702300
- [Derived] Weigert G, Kaya S, Pemp B, Sacu S, Lasta M, Werkmeister RM, Dragostinoff N, Simader C, Garhofer G, Schmidt-Erfurth U, Schmetterer L. Effects of lutein supplementation on macular pigment optical density and visual acuity in patients with age-related macular degeneration. Invest Ophthalmol Vis Sci. 2011 Oct 17;52(11):8174-8. doi: 10.1167/iovs.11-7522. PMID 21873668